CLINICAL TRIAL: NCT02681029
Title: Evaluating the Clinical Outcomes Following Transfer of Blastocysts Cultured From Thawed Cleavage Stage Embryos at Royan Institute: A Phase 3, Randomized Controlled Trial
Brief Title: The Clinical Outcomes Following Transfer of Blastocysts Cultured From Thawed Cleavage Stage Embryos
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Emb-023
Record Dates: First submitted 2016-02-02; First posted 2016-02-12 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2016-02

CONDITIONS: Infertility
Keywords: Cleavage stage blastocyst transfer cryopreservation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blastocyst transplantation (Experimental): The infertile women who underwent intra- uterus transferring of blastocyst from thawed cleavage embryo
  Interventions: Procedure: Blastocyte Transferring
- Control (Placebo Comparator): The infertile women who underwent intra- uterus transferring of thawed cleavage embryo.
  Interventions: Procedure: Embryo Transferring

INTERVENTIONS:
Procedure: Blastocyte Transferring — Intra-uterine transferring of blastocyst from thawed cleavage embryo in infertile women.
  Arms: Blastocyst transplantation
Procedure: Embryo Transferring — Inta-uterine transferring of thawed cleavage embryo transfer in infertile women.
  Arms: Control

SUMMARY:
Recent improvements in cell culture systems have led to a shift in in vitro fertilization (IVF) practice from early cleavage stage embryo transfer (ET) to blastocyst transfer. Blastocyst culture and transfer could theoretically provide better synchronization between the embryo and the uterine endometrium. The purpose of this study is comparing pregnancy rates and implantation rate following transfer of thawed cleavage embryos and blastocysts cultured from thawed cleavage embryos.

DETAILED DESCRIPTION:
The proposal of this study approved by our institutional review boards and institution's ethical committee, and all participants will sign a written consent before enter to study. All patients will be randomly divided into two groups of thawed cleavage embryo transfers and transfers of blastocysts from thawed cleavage embryos. Embryos will be transferred in hormone replacement cycles. Preparation of the endometrium will be started in the second day of menstruation and will be continued according to their transfer type (blastocyst or cleavage). βhCG will be assessed 14 days after embryo transfer. Treatment cycle outcomes will be compared between 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* The patients with first type of infertility
* Age ≤ 37 years
* Long ovulation induction protocol

Exclusion Criteria:

* Any previous surgery on the uterus and ovaries
* Uterine factor infertility
* Sever Male factor infertility (TESE, TESA ،Oligoteratozoospermia)
* Recurrent abortion
* The women with poor ovarian reserve

Ages: 16 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Actual)
Dates: Start 2015-11; Primary Completion 2020-07 (Actual); Study Completion 2020-09-27 (Actual)

PRIMARY OUTCOMES:
Pregnancy Rate | 4weeks
  Evaluation of pregnancy rate in women 4 weeks after embryos transfer (ET).

SECONDARY OUTCOMES:
Miscarriage Rate | 14 days
  Evaluation the miscarriage rate in women 14 days after embryo transfer (ET) with BHCG titration.
Implantation Rate | 14 days
  Evaluation the implantation rate in women 14 days after embryo transfer (ET) with BHCG titration..
Ongoing pregnancy rate | 14 days
  Evaluation the ongoing pregnancy rate in women 14 days after embryo transfer (ET) with BHCG titration..

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Tahereh Madani, MD, Study Director — Department of Endocrinology and Female Infertility, Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran; Poopak Eftekhari-Yazdi, PhD, Principal Investigator — Department of Endocrinology and Female Infertility, Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran; Nadia Jahangiri, MSc, Principal Investigator — Department of Endocrinology and Female Infertility, Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Madani T, Jahangiri N, Yahyaei A, Vesali S, Zarei M, Eftekhari-Yazdi P. Does The Culture of Post-Thawed Cleavage-Stage Embryos to Blastocysts Improve Infertility Treatment Outcomes of Frozen-Thawed Embryo Transfer Cycles? A Randomised Clinical Trial. Int J Fertil Steril. 2024 Feb 2;18(2):146-152. doi: 10.22074/ijfs.2023.560780.1357. PMID 38368518
- See also: Related Info — http://Royaninstitute.org